CLINICAL TRIAL: NCT04336267
Title: Anodal Transcranial Direct Current Stimulation in Chronic Migraine With and Medication Overuse Headache: a Pilot Randomized Sham-controlled Trial
Brief Title: Anodal tDCS in Chronic Migraine With Medication Overuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS-CM
Record Dates: First submitted 2020-03-28; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Chronic Migraine; Medication Overuse Headache
Keywords: Neuromodulation; Transcranial direct current stimulation; Chronic migraine; Medication overuse headache; EEG
MeSH Terms: conditions — Headache Disorders, Secondary | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Pilot randomized sham-controlled trial
Who Masked: Participant, Care Provider
Masking Description: Transcranial direct current stimulation (tDCS) was delivered by a technician that was not otherwise involved in the management of patients. The managing physician and the patient were instead blind to the type of stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcranial direct current stimulation (tDCS) group (Experimental): 7-day detoxification protocol + 5 consecutive days of anodal tDCS treatment over the primary motor cortex.
  Interventions: Device: Transcranial direct current stimulation (tDCS) group
- Sham group (Sham Comparator): 7-day detoxification protocol + 5 consecutive days of sham treatment over the primary motor cortex.
  Interventions: Device: Sham group

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) group — Patients randomized to the tDCS group were treated with the following parameters: duration of stimulation of 20 minutes per session with a 2 mA intensity of anodal stimulation.
  Arms: Transcranial direct current stimulation (tDCS) group
Device: Sham group — In the sham group, the stimulation setting was exactly the same but the stimulation intensity was set according to a ramping up/ramping down method and delivered only in the first and last 30 seconds of each session.
  Arms: Sham group

SUMMARY:
Non-invasive neuromodulation has been applied in several forms of primary headaches, and its usefulness has been suggested for both episodic and chronic migraine (CM). Transcranial direct current stimulation (tDCS) represents a non-invasive electrical stimulation technique that modulates neural brain activity by means of low amplitude direct current trough surface electrodes.

Very little evidence is available on the potential effect of tDCS in medication overuse and in the management of medication overuse headache (MOH), a condition frequently associated to CM.

CM associated to MOH still represents a challenge for physicians and patients due to the high prevalence in the general population, the associated severe disability, and the high costs imposed by the treatment.

The aim of the study was to investigate the possible application of tDCS in the management of CM associated to MOH. The primary objective of this pilot study was therefore to investigate the efficacy of anodal tDCS delivered on the primary motor cortex (M1) as add-on therapy to an in-hospital detoxification protocol in subjects affected by CM and MOH. The secondary objective was to evaluate the possible changes induced by tDCS on conventional EEG in order to obtain further clues about the effects of tDCS on brain activity.

DETAILED DESCRIPTION:
The study was a randomized, double-blind, controlled trial aimed at assessing the efficacy of five daily sessions of anodal t-DCS in add-on to a standardized in-hospital detoxification protocol in patients suffering from CM+MOH.

Twenty patients were enrolled among those consecutively attending the outpatient clinic of the IRCCS Mondino Foundation. All subjects underwent a screening visit with a physician of the Headache Science Centre of Mondino Institute. During the screening visit, a complete neurological and general examination was performed , and the inclusion/exclusion criteria were revised. Patients fulfilling criteria were enrolled in the baseline observation period for a month after an adequate training to monitor and record migraine and headache days, type and amount of acute medications and days of acute drug intake in an ad hoc diary. At the end of the baseline observation period, if inclusion/exclusion criteria were still satisfied, patients were randomized to the double-blind phase of the study (T0). To this end, patients were hospitalized on Mondays at the IRCCS Mondino Foundation for a 7-day detoxification protocol, that included: acute withdrawal of the overused drug and e.v. treatment with isotonic 0.9% NaCl saline 500 ml + cyanocobalamin 2500 mcg + folic acid 0.70 mg + nicotinamide 12 mg + ascorbic acid 150 mg + sodic glutathione 600 mg + delorazepam 0.5 mg administered b.i.d.

The day of hospital admission (T0), before the first infusion, patients were tested with a complete set of clinical scales and they completed the baseline EEG recording. After these procedures, the patients were randomized (1:1) to two different treatment groups: "tDCS group" or "sham group" and received 1 daily session of tDCS/sham stimulation for 5 consequent days (see below).

On day 5 (T1) patients underwent a follow-up EEG recording, administration of clinic scales for sleepiness, and attentional functions, evaluation of adverse events.

On day 7 patients were discharged from the hospital with or without the prescription of preventive medication (based on the physician judgement) and returned for a follow-up visit after 1 month (T2) and 6 months (T3). An addition EEG recording was obtained at T2.

Patients continued to record headache characteristic on the headache diary for the entire study observation period.

The study protocol was approved by the local Ethic Committee and all participants provided a written informed consent.

Transcranial direct current stimulation (tDCS) was delivered by a technician that was not otherwise involved in the management of patients. The managing physician were instead blind to the type of stimulation.

The technician used a specific battery-driven direct current stimulator (Newronika HDCstim, Newronika s.r.l.). The current was transferred by an approved saline-soaked pair of surface sponge electrodes (anode of 3x3 cm and cathode of 6x4 cm).

All the participants received daily stimulation sessions for 5 consecutive days (Monday to Friday). For the stimulation, the anode was placed over the primary motor cortex (M1), identified using the International 10-20 system for C3 (left M1) or C4 (right M1), and the cathode positioned over the contralateral supraorbital region (immediately below the Fp position of the 10-20 system). According to data from literature, in patients with a strict or prevalent (>70% of attacks) unilateral headache the contralateral hemisphere was stimulated, instead in patients with bilateral or shifting headache the dominant hemisphere was conventionally stimulated.

Patients randomized to the tDCS group were treated with the following parameters: duration of stimulation of 20 minutes per session with a 2 mA intensity of anodal stimulation.

In the sham group, the stimulation setting was exactly the same but the stimulation intensity was set according to a ramping up/ramping down method and delivered only in the first and last 30 seconds of each session. This stimulation paradigm is insufficient to produce a meaningful therapeutic effect, but it is necessary to guarantee to blind condition as it mimics the possible initial tingling sensation associated with active stimulation. All participants were informed about possible feelings related to tDCS treatment, such as a tingly sensation under the electrodes at the beginning of the stimulation. These procedures adequately blind participants to their group allocation. At the end of the 5 days stimulation period a blind check was performed.

An EEG recording was performed at baseline (T0), at the end of the tDCS/sham treatment (T1), and after 1 month from hospital discharge (T2).

The EEG was recorded with 19 Ag/AgCl electrodes which were placed according to the 10-20 EEG International System.

The EEG registration was performed in the morning (between 9:00 a.m. and 11 a.m.), in a dedicated sound-attenuated room by a technician blinded to the study procedures. The subjects were instructed to remain awake with their eyes closed. The EEG was recorded for 10 min with a sampling rate of 1024 Hz and it was filtered between 0.4 and 70 Hz. A Notch filter was also applied to avoid 50 Hz interferences.

For the EEG signal analysis, the investigators used a spectral analysis through a fast Fourier transformation. The investigators evaluated the power spectral density in these frequency ranges: Delta (1-4 Hz), Theta (4-8 Hz), Alpha (8-12 Hz), Beta (12-30 Hz). The absolute band power values (µV2) for each frequency were computed for each active electrode (Fp1, Fp2, F3, F4, F7, F8, Fz, C3, C4, Cz, P3, P4, Pz, T3, T4, T5, T6, O1, O2), using Cz as ground reference.

For statistical purpose, the band power values were expressed as the percentage variation respect to baseline (normalized as 100%). Moreover, in patients with tDCS/sham stimulation of the right hemisphere the investigators performed an offline virtual right to left inversion all the electrodes of the right hemisphere. In this setting, unless differently specified, all the odd electrodes were ipsilateral to the side of stimulation, while all the even electrodes were contralateral to the side of stimulation.

At T0 and T2 time points all patients completed a set of questionnaires to assess migraine-related disability, quality of life, sleep disturbances, and psychological aspects. The set included:

* the Migraine Disability Assessment (MIDAS) test;
* the Headache Impact Test-6 (HIT-6);
* Visual Analogue Scale (VAS);
* the Migraine-Specific Quality-of-Life Questionnaire (MSQ);
* Short Form Health Survey (SF-36);
* Sleep Condition Indicator (SCI);
* Pittsburgh Sleep Quality Index (PSQI);
* Zung scale for anxiety;
* Zung scale for depression.

Moreover, before every EEG recording (T0, T1, and T2), patients were tested for their level of sleepiness, and attentional functions with:

* Stanford Sleepiness Scale: 1-item questionnaire, with a score that range from 1 (optimal alertness) to 7 (high level of sleepiness);
* Symbol Digit Modalities Test (SDMT): the SDMT was administered to test attentive functions. Patients were trained to match numbers and abstract symbols, according to a coded key. The total score (0-110) is represented by the number of correct substitutions in 90 seconds, with higher values representative of better attention.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years;
* chronic migraine according to the criteria of the InternationaI Classification of Headache Disorders (code 1.3 ICHD-III) and Medication Overuse Headache (code 8.2 ICHD-III) present for at least 6 months at inclusion;
* previous failure of at least three prophylactic treatments.

Exclusion Criteria:

* other neurologic or neuropsychiatric diseases;
* other chronic painful syndromes;
* other types of primary or secondary headaches;
* use of a preventive medication at baseline;
* use of central nervous system modulating drugs;
* epilepsy;
* metallic head implants or use of a cardiac pacemaker;
* pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Headache frequency | Change in number of migraine days from T0 (baseline) to T2 (1 month after hospital discharge)
  Headache frequency measured by number of migraine days per month recorded in a headache diary.

SECONDARY OUTCOMES:
Migraine Disability Assessment (MIDAS) | Baseline (T0), after 1 month from hospital discharge (T2)
  Migraine related disability measured by the MIDAS. MIDAS test: 0-5 (grade I): minimal disability, 6-10 (grade II): mild disability, 11-20 (grade III): moderate disability, 21-40 (grade IVa): severe disability, 41 and higher (grade IVb): very severe disability.
Headache Impact Test-6 (HIT-6). | Baseline (T0), after 1 month from hospital discharge (T2)
  Migraine related disability measured by the HIT-6. A score of 49 or less: no impact, 50-55: some impact, 56-59: substantial impact, 60-78 severe impact.
Visual Analogue Scale (VAS) | Baseline (T0), after 1 month from hospital discharge (T2)
  Migraine related disability measured by VAS for pain intensity. VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Migraine-Specific Quality-of-Life Questionnaire (MSQ) | Baseline (T0), after 1 month from hospital discharge (T2)
  Migraine related disability measured by MSQ. It is a 14-item assessment, with each item rated on a 6-point scale (ranging from "none of the time" to "all of the time"). The investigators evaluated 3 scores, namely Role Function-Restrictive (RR), Role Function- Preventive (RP), and Emotional Function (EF). Raw scores have been transformed to a 100-point scale, with higher scores indicating better quality of life.
Short Form Health Survey (SF-36). | Baseline (T0), after 1 month from hospital discharge (T2)
  Migraine related disability measured by SF-36.It gives information about 8 different domains: physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items).
Sleep Condition Indicator (SCI) | Baseline (T0), after 1 month from hospital discharge (T2)
  Sleep quality measured by SCI. It is a 8-item questionnaire, with a score that range from 0 to 32. A higher score points toward a better sleep, while a score below 16 is significant for insomnia disorders.
Pittsburgh Sleep Quality Index (PSQI) | Baseline (T0), after 1 month from hospital discharge (T2)
  Sleep quality measured by PSQI. The questionnaire differentiates "poor" from "good" sleepers. A global score greater than five indicates poor sleep quality, with a maximum score of 21 (the worst overall sleep).
Zung scale for anxiety | Baseline (T0), after 1 month from hospital discharge (T2)
  Psychological aspects measured by the Zung scale for anxiety. It is a 20-item questionnaire, with a score that range from 20 to 80. A score above 36 is clinically significant for the presence of anxiety.
Zung scale for depression | Baseline (T0), after 1 month from hospital discharge (T2)
  Psychological aspects measured by the Zung scale for depression. It is a 20-item questionnaire with a score that range from 20 to 80. A score above 40 is clinically significant for the presence of depression.
EEG power spectrum (µV2) of alpha frequencies | Percentage modification of EEG power spectrum of alpha frequencies from T0 (baseline) to T2 (1 month after hospital discharge)
  For the EEG signal analysis, the investigators used a spectral analysis through a fast Fourier transformation. Epochs with eye movements, artifacts or periods of drowsiness were excluded from analysis. Power spectral density was calculated on the whole track, using a time windows of 5 seconds, with an overlapping of the samples equal to 50% and introducing zeropadding to reach a resolution of 0.1 Hz.
EEG power spectrum (µV2) of beta frequencies | Percentage modification of EEG power spectrum of beta frequencies from T0 (baseline) to T2 (1 month after hospital discharge)
  For the EEG signal analysis, the investigators used a spectral analysis through a fast Fourier transformation. Epochs with eye movements, artifacts or periods of drowsiness were excluded from analysis. Power spectral density was calculated on the whole track, using a time windows of 5 seconds, with an overlapping of the samples equal to 50% and introducing zeropadding to reach a resolution of 0.1 Hz.
EEG power spectrum (µV2) of theta frequencies | Percentage modification of EEG power spectrum of theta frequencies from T0 (baseline) to T2 (1 month after hospital discharge)
  For the EEG signal analysis, the investigators used a spectral analysis through a fast Fourier transformation. Epochs with eye movements, artifacts or periods of drowsiness were excluded from analysis. Power spectral density was calculated on the whole track, using a time windows of 5 seconds, with an overlapping of the samples equal to 50% and introducing zeropadding to reach a resolution of 0.1 Hz.
EEG power spectrum (µV2) of delta frequencies | Percentage modification of EEG power spectrum of delta frequencies from T0 (baseline) to T2 (1 month after hospital discharge)
  For the EEG signal analysis, the investigators used a spectral analysis through a fast Fourier transformation. Epochs with eye movements, artifacts or periods of drowsiness were excluded from analysis. Power spectral density was calculated on the whole track, using a time windows of 5 seconds, with an overlapping of the samples equal to 50% and introducing zeropadding to reach a resolution of 0.1 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, MD, Principal Investigator — IRCCS Mondino Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martelletti P, Jensen RH, Antal A, Arcioni R, Brighina F, de Tommaso M, Franzini A, Fontaine D, Heiland M, Jurgens TP, Leone M, Magis D, Paemeleire K, Palmisani S, Paulus W, May A; European Headache Federation. Neuromodulation of chronic headaches: position statement from the European Headache Federation. J Headache Pain. 2013 Oct 21;14(1):86. doi: 10.1186/1129-2377-14-86. PMID 24144382
- [Background] Palm U, Hasan A, Strube W, Padberg F. tDCS for the treatment of depression: a comprehensive review. Eur Arch Psychiatry Clin Neurosci. 2016 Dec;266(8):681-694. doi: 10.1007/s00406-016-0674-9. Epub 2016 Feb 3. PMID 26842422
- [Background] Solomons CD, Shanmugasundaram V. A review of transcranial electrical stimulation methods in stroke rehabilitation. Neurol India. 2019 Mar-Apr;67(2):417-423. doi: 10.4103/0028-3886.258057. PMID 31085852
- [Background] Feng Y, Zhang B, Zhang J, Yin Y. Effects of Non-invasive Brain Stimulation on Headache Intensity and Frequency of Headache Attacks in Patients With Migraine: A Systematic Review and Meta-Analysis. Headache. 2019 Oct;59(9):1436-1447. doi: 10.1111/head.13645. Epub 2019 Sep 18. PMID 31535368
- [Background] Dalla Volta G, Marceglia S, Zavarise P, Antonaci F. Cathodal tDCS Guided by Thermography as Adjunctive Therapy in Chronic Migraine Patients: A Sham-Controlled Pilot Study. Front Neurol. 2020 Feb 21;11:121. doi: 10.3389/fneur.2020.00121. eCollection 2020. PMID 32153497
- [Background] Westergaard ML, Glumer C, Hansen EH, Jensen RH. Prevalence of chronic headache with and without medication overuse: associations with socioeconomic position and physical and mental health status. Pain. 2014 Oct;155(10):2005-13. doi: 10.1016/j.pain.2014.07.002. Epub 2014 Jul 11. PMID 25020001
- [Background] Tassorelli C, Jensen R, Allena M, De Icco R, Sances G, Katsarava Z, Lainez M, Leston J, Fadic R, Spadafora S, Pagani M, Nappi G; the COMOESTAS Consortium. A consensus protocol for the management of medication-overuse headache: Evaluation in a multicentric, multinational study. Cephalalgia. 2014 Aug;34(9):645-655. doi: 10.1177/0333102414521508. Epub 2014 Feb 20. PMID 24558185
- [Background] Dasilva AF, Mendonca ME, Zaghi S, Lopes M, Dossantos MF, Spierings EL, Bajwa Z, Datta A, Bikson M, Fregni F. tDCS-induced analgesia and electrical fields in pain-related neural networks in chronic migraine. Headache. 2012 Sep;52(8):1283-95. doi: 10.1111/j.1526-4610.2012.02141.x. Epub 2012 Apr 18. PMID 22512348
- [Background] Auvichayapat P, Janyacharoen T, Rotenberg A, Tiamkao S, Krisanaprakornkit T, Sinawat S, Punjaruk W, Thinkhamrop B, Auvichayapat N. Migraine prophylaxis by anodal transcranial direct current stimulation, a randomized, placebo-controlled trial. J Med Assoc Thai. 2012 Aug;95(8):1003-12. PMID 23061303
- [Background] Przeklasa-Muszynska A, Kocot-Kepska M, Dobrogowski J, Wiatr M, Mika J. Transcranial direct current stimulation (tDCS) and its influence on analgesics effectiveness in patients suffering from migraine headache. Pharmacol Rep. 2017 Aug;69(4):714-721. doi: 10.1016/j.pharep.2017.02.019. Epub 2017 Mar 1. PMID 28551531
- [Background] Lewis GN, Rice DA, Kluger M, McNair PJ. Transcranial direct current stimulation for upper limb neuropathic pain: A double-blind randomized controlled trial. Eur J Pain. 2018 Aug;22(7):1312-1320. doi: 10.1002/ejp.1220. Epub 2018 Apr 17. PMID 29577496
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] Espie CA, Farias Machado P, Carl JR, Kyle SD, Cape J, Siriwardena AN, Luik AI. The Sleep Condition Indicator: reference values derived from a sample of 200 000 adults. J Sleep Res. 2018 Jun;27(3):e12643. doi: 10.1111/jsr.12643. Epub 2017 Nov 29. PMID 29193493
- [Background] Fellows RP, Schmitter-Edgecombe M. Symbol Digit Modalities Test: Regression-Based Normative Data and Clinical Utility. Arch Clin Neuropsychol. 2019 Jan 24;35(1):105-115. doi: 10.1093/arclin/acz020. PMID 31329813
- [Background] Pijpers JA, Kies DA, Louter MA, van Zwet EW, Ferrari MD, Terwindt GM. Acute withdrawal and botulinum toxin A in chronic migraine with medication overuse: a double-blind randomized controlled trial. Brain. 2019 May 1;142(5):1203-1214. doi: 10.1093/brain/awz052. PMID 30982843
- [Background] Tassorelli C, Jensen R, Allena M, De Icco R, Katsarava Z, Miguel Lainez J, Leston JA, Fadic R, Spadafora S, Pagani M, Nappi G; COMOESTAS Consortium. The added value of an electronic monitoring and alerting system in the management of medication-overuse headache: A controlled multicentre study. Cephalalgia. 2017 Oct;37(12):1115-1125. doi: 10.1177/0333102416660549. Epub 2016 Jul 20. PMID 27440251
- [Background] Nielsen M, Carlsen LN, Munksgaard SB, Engelstoft IMS, Jensen RH, Bendtsen L. Complete withdrawal is the most effective approach to reduce disability in patients with medication-overuse headache: A randomized controlled open-label trial. Cephalalgia. 2019 Jun;39(7):863-872. doi: 10.1177/0333102419828994. Epub 2019 Feb 7. PMID 30732459
- [Background] Andrade SM, de Brito Aranha REL, de Oliveira EA, de Mendonca CTPL, Martins WKN, Alves NT, Fernandez-Calvo B. Transcranial direct current stimulation over the primary motor vs prefrontal cortex in refractory chronic migraine: A pilot randomized controlled trial. J Neurol Sci. 2017 Jul 15;378:225-232. doi: 10.1016/j.jns.2017.05.007. Epub 2017 May 3. PMID 28566169
- [Background] Rocha S, Melo L, Boudoux C, Foerster A, Araujo D, Monte-Silva K. Transcranial direct current stimulation in the prophylactic treatment of migraine based on interictal visual cortex excitability abnormalities: A pilot randomized controlled trial. J Neurol Sci. 2015 Feb 15;349(1-2):33-9. doi: 10.1016/j.jns.2014.12.018. Epub 2014 Dec 18. PMID 25579414
- [Background] Tassorelli C, Diener HC, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of chronic migraine in adults. Cephalalgia. 2018 Apr;38(5):815-832. doi: 10.1177/0333102418758283. Epub 2018 Mar 4. PMID 29504482
- [Background] Granato A, Fantini J, Monti F, Furlanis G, Musho Ilbeh S, Semenic M, Manganotti P. Dramatic placebo effect of high frequency repetitive TMS in treatment of chronic migraine and medication overuse headache. J Clin Neurosci. 2019 Feb;60:96-100. doi: 10.1016/j.jocn.2018.09.021. Epub 2018 Oct 11. PMID 30316627
- [Background] Coppola G, Di Lorenzo C, Parisi V, Lisicki M, Serrao M, Pierelli F. Clinical neurophysiology of migraine with aura. J Headache Pain. 2019 Apr 29;20(1):42. doi: 10.1186/s10194-019-0997-9. PMID 31035929
- [Background] De Pascalis V, Scacchia P. The influence of reward sensitivity, heart rate dynamics and EEG-delta activity on placebo analgesia. Behav Brain Res. 2019 Feb 1;359:320-332. doi: 10.1016/j.bbr.2018.11.014. Epub 2018 Nov 12. PMID 30439452
- [Background] Porcaro C, Di Lorenzo G, Seri S, Pierelli F, Tecchio F, Coppola G. Impaired brainstem and thalamic high-frequency oscillatory EEG activity in migraine between attacks. Cephalalgia. 2017 Sep;37(10):915-926. doi: 10.1177/0333102416657146. Epub 2016 Jun 29. PMID 27358281
- [Background] Hodkinson DJ, Wilcox SL, Veggeberg R, Noseda R, Burstein R, Borsook D, Becerra L. Increased Amplitude of Thalamocortical Low-Frequency Oscillations in Patients with Migraine. J Neurosci. 2016 Jul 27;36(30):8026-36. doi: 10.1523/JNEUROSCI.1038-16.2016. PMID 27466345